CLINICAL TRIAL: NCT03595267
Title: Optimal Approaches to Chronic Kidney Disease Case Finding in Indigenous Communities
Brief Title: Kidney Check: Diabetes, Blood Pressure & Kidney Health Checks & Care in Indigenous Communities.
Status: Recruiting | Type: Observational
Sponsor: University of Manitoba (Other)
Collaborators: Canadians Seeking Solutions and Innovations to Overcome Chronic Kidney Disease (Other); Alberta Health services (Other); First Nations Health Authority (Unknown); First Nations Health and Social Secretariat of Manitoba (Unknown); Research Manitoba (Other); Shared Health Laboratory Services of Manitoba (Unknown); Seven Oaks Hospital Chronic Disease Innovation Centre Inc. (Unknown); Keewatinohk Inniniw Minoayawin Inc. (KIM) (Unknown)
Responsible Party: Principal Investigator, Dr. Paul Komenda, Professor, University of Manitoba
Other Study IDs: HS20110 (H2016:348)
Record Dates: First submitted 2018-07-12; First posted 2018-07-23 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Chronic Kidney Disease; Diabetes; Hypertension
Keywords: Indigenous Canadians; Screening Study
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus; Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rural and Remote Indigenous Communities: Point-of-care screening for Chronic Kidney Disease, Diabetes, and Hypertension will be administered in rural and remote communities in Manitoba, British Columbia, Alberta, Saskatchewan, and Ontario.
  Interventions: Other: Point-of-care screening

INTERVENTIONS:
Other: Point-of-care screening — After consent is obtained, a registered nurse will administer a demographic questionnaire, collecting the participant's personal health number, age, gender, date of birth, and name of community. Physical data including height, weight, and blood pressure will also be collected. A blood sample and a urine sample will be taken, with point-of-care testing being performed during the screening appointment to allow for results of the testing to be received and discussed with each patient at the time of the appointment. After screening, to ensure a "closed loop" system of care, patients at the highest risk of kidney failure will be referred to a nephrologist, while those at lower risk will be referred to their primary care provider with specific treatment and re-testing recommendations.

SUMMARY:
Faced with limited access to preventative health care services, Indigenous people living in rural and remote communities are at a higher risk of Chronic Kidney Disease (CKD) and kidney failure, when compared to the general population. The goal of this project is to perform point-of-care testing for CKD and its risk factors, including diabetes and high blood pressure, for individuals residing in rural and remote Indigenous communities across the Canadian provinces of Manitoba, British Columbia, Alberta, Saskatchewan, and Ontario. In addition to providing individuals with information about their risk of developing CKD, as well as providing tailored treatment plans, this study will help provide evidence to develop a permanent CKD surveillance system in all Indigenous communities across Canada, consequently decreasing the burden of CKD and kidney failure in these communities.

DETAILED DESCRIPTION:
Compared to the general population, Indigenous people disproportionately suffer from higher rates of diabetes, hypertension, obesity, and chronic kidney disease (CKD), when compared to their non-Indigenous counterparts. However, rates of these morbidities are greatest for Indigenous individuals living in rural and remote areas, where social inequalities such as poverty and poor access to services - in particular reduced access to primary care and nephrology specialists - are the most the salient.

If caught and treated early in its course, kidney failure is often preventable, especially for those at the highest risk of progression. However, CKD is often unrecognizable and asymptomatic until it is in its later stages, when the chances of preventing kidney failure are limited. Therefore, in order to administer targeted therapeutic interventions, early identification and stratification of those at highest risk of CKD are urgently needed. Screening programs using state of the art point-of-care testing equipment with blood and urine samples can test for CKD both quickly and accurately. While general population-based screening have not been found to be beneficial, targeted screening directed toward high-risk patients with diabetes and high blood pressure, or high-risk populations known to progress rapidly or have limited access to primary health care, are cost-effective. In particular, research has shown that the cost utility of one-off, point-of-care screening and treatment for CKD in rural and remote Indigenous communities is highly cost-effective when compared to usual care provided in these geographic areas.

The goal of this project is to develop a platform that will enable the early diagnosis of Indigenous adults and children with CKD living in Indigenous communities across Canada, and lead to treatment and follow up care targeted to each individual's risk of kidney failure. By developing mobile mass screening and prevention initiatives in adults and children for the prevention of CKD and kidney failure, appropriate treatment and follow-up will continue, and rates of CKD progression will decline, with fewer patients reaching kidney failure requiring dialysis. In addition, this project will further demonstrate the benefits of front line surveillance, risk prediction and treatment, and lead to novel insights regarding prognosis, and the factors driving kidney disease in Indigenous communities, ultimately serving as the gold-standard model for delivery of kidney care across Canada.

ELIGIBILITY:
Inclusion Criteria:

* All individuals aged 10 years old - 80 years old will be recruited for screening, regardless of known CKD risk factors, such as diabetes, elevated blood pressure, or family history of kidney disease.

Exclusion Criteria:

* None.

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Indigenous communities in rural (accessible by road), and remote (accessible by flying-in, or winter ice roads) areas of Manitoba, British Columbia, Alberta, Saskatchewan and Ontario will be targeted for the screening program.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Biomarkers of Kidney Function | 1 day (At time of screening)
  eGFR; Albuminuria; Urine ACR
Diabetes | 1 day (At time of screening)
  Defined as a Hemoglobin A1c => 6.5%
Elevated Blood Pressure | 1 day (At time of screening)
  Defined as a Systolic Blood Pressure > 140 mmHg, or Diastolic Blood Pressure > 90mmHg
Kidney Failure Risk | 1 day (At time of screening)
  Measured using the Kidney Failure Risk Equation

CONTACTS AND LOCATIONS:
Overall Officials: Paul Komenda, MD MHA, Principal Investigator — University of Manitoba
Locations (3):
- Canada (3):
  - Alberta Health Services, Calgary, Alberta
  - First Nations Research and Knowledge Exchange, West Vancouver, British Columbia
  - Chronic Disease Innovation Centre, Winnipeg, Manitoba

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lavallee B, Chartrand C, McLeod L, Rigatto C, Tangri N, Dart A, Gordon A, Ophey S, Komenda P. Mass screening for chronic kidney disease in rural and remote Canadian first nations people: methodology and demographic characteristics. Can J Kidney Health Dis. 2015 Mar 19;2:9. doi: 10.1186/s40697-015-0046-9. eCollection 2015. PMID 27408755
- [Background] Komenda P, Lavallee B, Ferguson TW, Tangri N, Chartrand C, McLeod L, Gordon A, Dart A, Rigatto C. The Prevalence of CKD in Rural Canadian Indigenous Peoples: Results From the First Nations Community Based Screening to Improve Kidney Health and Prevent Dialysis (FINISHED) Screen, Triage, and Treat Program. Am J Kidney Dis. 2016 Oct;68(4):582-590. doi: 10.1053/j.ajkd.2016.04.014. Epub 2016 May 30. PMID 27257016
- [Background] Ferguson TW, Tangri N, Tan Z, James MT, Lavallee BDA, Chartrand CD, McLeod LL, Dart AB, Rigatto C, Komenda PVJ. Screening for chronic kidney disease in Canadian indigenous peoples is cost-effective. Kidney Int. 2017 Jul;92(1):192-200. doi: 10.1016/j.kint.2017.02.022. Epub 2017 Apr 20. PMID 28433383
- [Background] Harasemiw O, Milks S, Oakley L, Lavallee B, Chartrand C, McLeod L, Di Nella M, Rigatto C, Tangri N, Ferguson T, Komenda P. Remote Dwelling Location Is a Risk Factor for CKD Among Indigenous Canadians. Kidney Int Rep. 2018 Feb 10;3(4):825-832. doi: 10.1016/j.ekir.2018.02.002. eCollection 2018 Jul. PMID 29989009
- [Background] Komenda P, Ferguson TW, Macdonald K, Rigatto C, Koolage C, Sood MM, Tangri N. Cost-effectiveness of primary screening for CKD: a systematic review. Am J Kidney Dis. 2014 May;63(5):789-97. doi: 10.1053/j.ajkd.2013.12.012. Epub 2014 Feb 12. PMID 24529536
- [Background] Dart A, Lavallee B, Chartrand C, McLeod L, Ferguson TW, Tangri N, Gordon A, Blydt-Hansen T, Rigatto C, Komenda P. Screening for kidney disease in Indigenous Canadian children: The FINISHED screen, triage and treat program. Paediatr Child Health. 2018 Nov;23(7):e134-e142. doi: 10.1093/pch/pxy013. Epub 2018 Apr 14. PMID 30374222
- [Background] Curtis S, Martin H, DiNella M, Lavallee B, Chartrand C, McLeod L, Woods C, Dart A, Tangri N, Rigatto C, Komenda P. Kidney Check Point-of-Care Testing-Furthering Patient Engagement and Patient-Centered Care in Canada's Rural and Remote Indigenous Communities: Program Report. Can J Kidney Health Dis. 2021 Mar 31;8:20543581211003744. doi: 10.1177/20543581211003744. eCollection 2021. PMID 33868690
- [Background] Curtis S, Sokoro A, Martin H, McLeod L, Chartrand C, Lavallee B, Woods C, Di Nella M, Levin A, Komenda P. A Comprehensive Quality Assurance Platform in Canada for National Point-of-Care Chronic Kidney Disease Screening: The Kidney Check Program. Kidney Int Rep. 2020 Dec 30;6(2):513-517. doi: 10.1016/j.ekir.2020.11.031. eCollection 2021 Feb. No abstract available. PMID 33615077
- See also: Study website — http://kidneycheck.ca